CLINICAL TRIAL: NCT02605629
Title: EValuation of the Impact of a TOpical Lotion, CG428, on Permanent Chemotherapy Induced Hair and Scalp Disorders in Cancer SUrvivors: A randoMized, Single-center, Double-blind placEbo Controlled Trial (a Pilot Study)
Brief Title: EValuation of the Impact of a TOpical Lotion on Permanent Chemotherapy Induced Hair Disorders in Cancer Survivors
Acronym: VOLUME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Legacy Healthcare Services (Other)
Responsible Party: Principal Investigator, Juhee Cho, Cancer Education Center, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VOLUME
Record Dates: First submitted 2015-11-10; First posted 2015-11-16 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia | interventions — CG428

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CG428 (Experimental): Patients will self-administer the study product twice per day (morning, evening) for 6 months, for the efficacy assessment
  Interventions: Other: CG428
- Placebo (Placebo Comparator): Patients will self-administer the study placebo twice per day (morning, evening) for 6 months, for the efficacy assessment
  Interventions: Other: Placebo

INTERVENTIONS:
Other: CG428 — The experimental group will receive CG428. For each application, the patient should shake the bottle before spraying 10-12 times directly to the dry scalp whole area, with the nozzle, and then gently massage the whole scalp with fingertips in order to spread the lotion evenly until it has completely penetrated the scalp. Hairs should not be washed or shampooed within 1 hour following study treatment administration. Each dose should be spaced out by minimum 4 hours.
  Arms: CG428
Other: Placebo — The placebo group will received placebo which excluded active ingredients. For each application, the patient should shake the bottle before spraying 10-12 times directly to the dry scalp whole area, with the nozzle, and then gently massage the whole scalp with fingertips in order to spread the lotion evenly until it has completely penetrated the scalp. Hairs should not be washed or shampooed within 1 hour following study treatment administration. Each dose should be spaced out by minimum 4 hours.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the Impact of a topical Lotion, CG428, on permanent chemotherapy induced hair and scalp disorders in Cancer survivors. This is a double-blind, single center, randomized, controlled trial in breast cancer survivors.

Hair condition and parameters of 61 breast cancer survivors who were previously included in DERMA study (a prospective cohort study to assess appearance changes due to breast cancer treatment completed in July, 13th,2013) will be assessed.

1. Patients whose hair parameters are below the baseline as measured before the start of the chemotherapy or
2. who complain from incomplete hair regrowth will be eligible to participate in the randomized controlled trial.

Patients who agree to participant in the study will be randomly assigned to two parallel arms (Arm 1: CG428/ Arm 2: Placebo). Patients will self-administer the study product or placebo twice per day (morning, evening) for 6 months, for the efficacy assessment.

Primary endpoint was recovery of hair thickness 6 months after intervention as assessed using Folliscope 4.0.

Secondary endpoints included hair density at 6 months after intervention, distress due to chemotherapy induced alopecia, scalp skin parameters (water and sebum). Patient-reported hair quality improvement, body image and quality of life, and time to first visible improvement based on global photographs of hair and nails.

DETAILED DESCRIPTION:
The research team at Cancer Education Center at Samsung Comprehensive Cancer Center has studied CIA and its impact on distress and psychosocial well-being since 2008. We found that more than half of the breast cancer patients experienced higher distress due to CIA, during cancer treatment, and this distress was strongly associated with negative body image, overall health status, and psychosocial well-being. In a recent prospective cohort study, we assessed skin and hair change patterns before, during and 6 months after chemotherapy in 61 volunteers. We found that the majority of the patients still experienced CIA at 6 months after completion of chemotherapy. Actually, hair diameter at 6th month after chemotherapy had not recovered to baseline level. Permanent chemotherapy-induced alopecia, defined as absent or incomplete hair regrowth at ≥6 months post-chemotherapy, was reported from 53 to 74%. Like CIA, permanent CIA also lacks recognition and has been underserved regardless of patients' needs. The first botanical blend Legacy Healthcare developed and patented is Cellium. Cellium is composed of 4 botanicals (Allium cepa L., Citrus limon L., Theobroma cacao L., Paullinia cupana). The first product derived from Cellium is a topical lotion for male and female alopecia, CG210. Based on the safety and efficacy data, the EMA (European Medicines Agency) has considered CG210 eligible for a European centralized herbal medicine registration. CG428 is the second product derived from Cellium. CG428 contains the exact same ingredients as CG210, in a different dosage. Legacy Healthcare have conducted a pilot studies with CG428 in Japan. The trial included female cancer survivors experiencing permanent/persistent CIA for more than 12. Based on the results, several cancer treatment centers in Japan have started to recommend the product on a compassionate basis.We therefore hypothesize that the investigated topical lotion may mitigate the impact of protracted or permanent CIA in cancer survivors by restoring a normalized apoptotic process of hair follicular cells and reducing the acute, as well as chronic inflammation in the scalp, two issues that may remain unsettled following anticancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* hair parameters obtained before the start of chemotherapy
* hair parameters obtained 6 months after the completion of chemotherapy

  * whose hair parameters are below the baseline, as measured before the start of chemotherapy during DERMA study, or
  * who complain from incomplete hair regrowth at the time of enrollment (on average 24 months after chemotherapy completion)
* Able to keep their hair style

  * Able to use the study treatment in compliance with the protocol.
* Physical (ECOG≤1) and psychological ability to participate

Exclusion Criteria:

* Concomitant use of other anti-hair-loss treatment or hair growth treatment.
* Patients with recent hair transplants or who plan to have transplants.
* Known allergy or hypersensitivity to some components of CG428 (including allium cepa (onion), citrus, caffeine, the obromine)
* Pre-existing alopecia or significant scalp disease, which may alter study treatment administration or absorption.

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
Recovery rate of hair thickness 6 months after intervention Using Folliscope 4.0, LeadM | 6 months after randomization
  Objectively quantified hair thickness will measure using Folliscope 4.0, LeadM We will take a picture of 15X and 60X on the parietal (To around 2 cm) and then analysis using Folliscope program.

SECONDARY OUTCOMES:
Chemotherapy-induced alopecia distress Stress Using Chemotherapy induced alopecia distress scale (CADS) | 6 months after randomization
  Respondents will be instructed to indicate on a 4-point Likert scale on each statement (1=Not at all, 2= A little, 3=Quite a bit, 4=Very much). Total scores will be calculated by summing responses for all items; higher scores means more distress due to CIA
Global photographs | All time (baseline, 3month and 6 months after intervention)
  Pictures to be focused on head/hair, which means shorter distance between the equipment and the subject using Canon EOS 70D
Scalp skin water levels | All time (baseline, 3month and 6 months after intervention)
  Water on scalp: it will be measured using Corneometer (Courage-Khazakaelectronic GmbH, Germany). We will measure 3 times on same area
Sebum on scalp | All time (baseline, 3month and 6 months after intervention)
  it will be measured using Sebumeter SM815 (Courage-Khazakaelectronic GmbH, Germany). We will measure 1 times on same area
Overall hair and scalp condition | All time (baseline, 3month and 6 months after intervention)
  Patient self-assessment: We will measure patient reported hair density and thickness, scalp condition, and density using visual analogue scale (VAS) ranging from 0 to 10
Nail condition | All time (baseline, 3month and 6 months after intervention)
  Patient self-assessment: We will use self-reported questionnaire using visual analogue scale (VAS) ranging from 0 to 10.
  Global photographs: We will take a picture the patients' nail using Canon EOS 70D with Intelli-Flash system or similar system
Quality of life at the time | All time (baseline, 3month and 6 months after intervention)
  We will assess patients' body image using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 and breast specific module
Depression | All time (baseline, 3month and 6 months after intervention)
  We will assess patients' depression using Hospital Anxiety and Depression Scale (HADS). It consists of 14 items in two domains (Depression and anxiety).
Anxiety | All time (baseline, 3month and 6 months after intervention)
  We will assess patients' anxiety using Hospital Anxiety and Depression Scale (HADS). It consists of 14 items in two domains (Depression and anxiety).
Satisfaction with products | After intervention (3month and 6 months after intervention)
  We will use self-reported questionnaire for satisfaction with the products as well as suggestions for improvement after completion of study with patients who received the CG428.
Hair condition | All time (baseline, 3month and 6 months after intervention)
  Outcomes will be collected using objective methods and patient reported outcomes:
  Objectively quantified: Hair thickness and density: We will measure hair thickness and density using Folliscope 4.0, LeadM We will take a picture on the parietal (To around 2 cm) and then analysis using Folliscope program.
  Global photographs: Pictures to be focused on head/hair, which means shorter distance between the equipment and the subject

OTHER OUTCOMES:
Effort for managing hair | All time (baseline, 3month and 6 months after intervention)
  Effort for managing hair using a questionniare whcih developed by researcher

CONTACTS AND LOCATIONS:
Overall Officials: Juhee Cho, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Danbee Kang, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim IR, Cho J, Choi EK, Kwon IG, Sung YH, Lee JE, Nam SJ, Yang JH. Perception, attitudes, preparedness and experience of chemotherapy-induced alopecia among breast cancer patients: a qualitative study. Asian Pac J Cancer Prev. 2012;13(4):1383-8. doi: 10.7314/apjcp.2012.13.4.1383. PMID 22799336
- [Background] Choi EK, Kim IR, Chang O, Kang D, Nam SJ, Lee JE, Lee SK, Im YH, Park YH, Yang JH, Cho J. Impact of chemotherapy-induced alopecia distress on body image, psychosocial well-being, and depression in breast cancer patients. Psychooncology. 2014 Oct;23(10):1103-10. doi: 10.1002/pon.3531. Epub 2014 Mar 24. PMID 24664939
- [Background] Kang D, Kim IR, Im YH, Park YH, Ahn JS, Lee JE, Nam SJ, Park H, Kim E, Lee HK, Lee DY, Cho J. Quantitative changes in skin composition parameters due to chemotherapy in breast cancer patients: a cohort study. Breast Cancer Res Treat. 2015 Aug;152(3):675-82. doi: 10.1007/s10549-015-3502-4. Epub 2015 Jul 22. PMID 26198993
- [Background] Kondo R et al.,Assessment of the Efficacy of CG 428 in the Recovery from Chemotherapy Long Term Side Effects on Hair in Women (an open label evaluation), Legacy Healthcare Japan, 2013